CLINICAL TRIAL: NCT02219139
Title: A Comparative, Randomized, Prospective, Clinical Pilot Study to Evaluate the Performance of Modified Study Abutments in Single Tooth Gaps
Brief Title: A Comparative, Randomized, Prospective, Performance Evaluation of Abutments in Single Tooth Gaps
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients could be recruited
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CR 03/10 ESTA; CIV-12-10-009101 (Other: EUDAMED)
Record Dates: First submitted 2014-07-17; First posted 2014-08-18 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Tooth Loss
Keywords: Edentulous; Roxolid; SLAclive surface; Titanium/zirconium
MeSH Terms: conditions — Tooth Loss; Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ESTA abutment Roxolid (Other): One study abutment per patient will be placed. After healing for 6 to 7 weeks, patients will be asked to stop oral hygiene at the study site for 2 weeks.
  Sulcus fluid and plaque samples will be taken at the abutment site at several visits before and during abdication of oral hygiene.
  The study finishes with biopsy visit. Afterwards a regular abutment will be placed and the patients will be treated according to the standard protocol of the clinic to obtain their final restoration.
  Interventions: Device: ESTA abutment Roxolid

INTERVENTIONS:
Device: ESTA abutment Roxolid — Enhanced Soft Tissue Attachment surface on Roxolid or machined surface on Roxolid abutment placement.

SUMMARY:
Immunologically evaluation of myeloperoxidase level as indicator for inflammatory reactions on modified surface abutments compared to machined surface abutments.

DETAILED DESCRIPTION:
One study abutment per patient will be placed. After healing for 6 to 7 weeks, patients will be asked to stop oral hygiene at the study site for 2 weeks.

Sulcus fluid and plaque samples will be taken at the abutment site at several visits before and during abdication of oral hygiene.

The study finishes with biopsy visit. Afterwards a regular abutment will be placed and the patients will be treated according to the standard protocol of the clinic to obtain their final restoration

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have voluntary signed the informed consent form before any study related action.
* Males and females with at least 18 years of age
* Non-smokers
* Straumann bone level implant (healed for at least 4 weeks) in a tooth gap in the maxilla or mandible with thick tissue biotype
* Adequate oral hygiene (Full mouth plaque index; O'Leary, et al. 1972) <25% at abutment placement
* The patient must be able to open the mouth to allow removal of the abutment at the planned abutment site

Exclusion Criteria:

* Systemic disease that would interfere with dental implant therapy (e.g. uncontrolled diabetes)
* Any antibiotic treatment or anti-inflammatory treatment within the past 2 month
* Any contraindications for oral surgical procedures
* Mucosal diseases (e.g. lichen planus, mouth ulcer)
* History of local irradiation therapy
* Current treated (within the last 12 month) or untreated periodontitis
* Current treated (within the last 6 month) or untreated gingivitis
* Probing pocket depth of ≥4 mm on one of the teeth immediately adjacent to the dental implant site
* Severe bruxing or clenching habits
* Lack of primary stability of the implant at abutment placement
* Subjects who have undergone administration of any investigational device within 30 days of enrolment in the study
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance or unreliability
* Physical or mental handicaps that would interfere with the ability to follow protocol procedures
* Pregnant or breastfeeding wome
* Insufficient soft tissue attachment to the neck of the abutment (e.g. visibility of the abutment platform or exposed ESTAnsurface) after abutment placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Myeloperoxidase level as indicator for inflammatory reactions on modified surface abutments compared to machined surface abutments. | Inflammation assessment and biopsy at study day 70.
  A biopsy will be taken at study day 70. The study abutment will be removed together with a small slice of the surrounding soft tissue to histologically evaluation.

SECONDARY OUTCOMES:
Evaluation of myeloperoxidase level of modified surface abutments compared to machined surface abutment at visit 2, 3, 4, and 6. | 20-24 weeks
  A immunology sample will be taken 2-3 weeks after abutment placement, followed on week 6-7, week 8, week 9, and at week 20-24.
evaluation of inflammatory parameters of modified surface abutment compared to machined surface abutments | 20-24 weeks
  A immunology sample will be taken 2-3 weeks after abutment placement, followed on week 6-7, week 8, week 9, and at week 20-24.
Evaluation of clinical inflammatory parameters of modified surface abutments compared to machined surface abutments based on modified Mombelli plaque index and modified Lobene gingival index. | 20-24 weeks
  A immunology sample will be taken 2-3 weeks after abutment placement, followed on week 6-7, week 8, week 9, and at week 20-24.
Evaluation of subgingival plaque extension of modified surface abutments compared to machined surface abutments | 9 weeks after abutment placement
  Patients will be asked to suspend oral hygiene in the area of the abutment. after 42-49 days after abutment placement for 14 days. At study week 8 a histological sample will be taken
Evaluation of soft tissue around the abutment of modified surface abutment compared to machined surface abutments | At 8 weeks after abutment placement
  8 weeks after abutment placement patients have been asked for 14 days of abdication of oral hygiene. A histological sample will be taken then.
Evaluation of bacterial community at the abutment site | 28 days
  At study day 42-49, day 49-56, day 56-63, and day 77-105 a microbiological sample will be taken

CONTACTS AND LOCATIONS:
Overall Officials: Anton Sculean, Dr med dent, Principal Investigator — University Bern, Zahnmedizinische Kliniken Bern
Locations (1):
- Universität Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No